CLINICAL TRIAL: NCT06797375
Title: Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RLYB116 in Healthy Participants
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of RLYB116 in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rallybio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPC2401
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hematologic Diseases; Autoimmune Diseases
Keywords: complement-mediated diseases
MeSH Terms: conditions — Hematologic Diseases; Autoimmune Diseases | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- RLYB116 Dose 1 (Experimental): RLYB116 for Injection Dose 1, weekly for 5 weeks
  Interventions: Drug: RLYB116 for Injection
- RLYB116 Dose 2 (Experimental): RLYB116 for Injection Dose 2, weekly for 5 weeks
  Interventions: Drug: RLYB116 for Injection
- Placebo for Injection (Placebo Comparator): Sodium chloride injection, 0.9% saline (for both RLYB116 doses), weekly for 5 weeks
  Interventions: Drug: RLYB116 for Injection

INTERVENTIONS:
Drug: RLYB116 for Injection — RLYB116 is a small protein composed of an Affibody® Z-domain that binds with high affinity to C5, inhibiting terminal complement activation, and an albumin binding domain (ABD) that extends the effective plasma half-life of the protein by targeting serum albumin.

SUMMARY:
This study will investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of RLYB116 (with an improved impurity profile) following repeated administration of RLYB116 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants, 18 to 55 years of age.
2. Able to provide written informed consent.
3. Body mass index (BMI) of 18.0 to 32.0 kg/m2.
4. Must have been vaccinated against N. meningitidis and S. pneumoniae with approved vaccine according to product label. All participants considered eligible for enrollment will be vaccinated or willing to receive vaccination according to the following:

   1. Vaccination with Meningococcal Group A, C, W135, and Y conjugate vaccine (Menveo® or an acceptable alternative) + Pneumococcal Polysaccharide Vaccine (Pneumovax® 23 or an acceptable alternative) at least 28 days prior to receiving the first dose of RLYB116.
   2. Vaccination with Meningococcal Group B (Bexsero®) at least 14 days prior to receiving the first dose of RLYB116.

Exclusion Criteria:

1. Participants that smoke more than 10 cigarettes per week
2. Positive serology for HIV or active infection with hepatitis B virus or hepatitis C virus.
3. Pregnant or nursing
4. Donation or loss of greater than 400 mL of blood within 56 days of study enrollment
5. History of severe hypersensitivity to any drug, including penicillin or ciprofloxacin, or to N. meningitidis or S. pneumoniae vaccines.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as defined by CTCAE 5.0. | From baseline to Day 1, 2, 3, 4, 5, 8, 9, 15, 16, 22, 23, 29, 30, 32, 33, 36, 43, 57, 71, 99

SECONDARY OUTCOMES:
Inhibition of complement activation measured by free/total C5 concentrations and hemolytic activity | Day 1, 2, 8, 15, 29, 20, 32, 33, 43, 57, 71, 99
Anti-RLYB116 antibodies measured in serum | Day 1, 29, 99
Exposure to RLYB116 as measured in serum | Day 1, 2, 3, 4, 5, 8, 15, 29, 53, 57, 71, 99

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Brisbane, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No